CLINICAL TRIAL: NCT03218644
Title: Effectiveness of a Propioceptive Exercise Program in Subjects With Inespecific Neck Pain
Brief Title: Effectiveness of Proprioceptive Exercise in Neck Pain
Acronym: PropNeckPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID0017
Record Dates: First submitted 2017-07-08; First posted 2017-07-14 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Neck Pain
Keywords: Proprioception
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Follow the usual treatment and perform the exercises of cervical mobility before a mirror.
  Interventions: Other: Mobility exercises
- Experimental group (Experimental): The same procedure is followed by substituting proprioceptive exercises for craniocervical sensorimotor control with a laser instrument located on the patient's head and a target.
  Interventions: Other: Proprioception exercises

INTERVENTIONS:
Other: Mobility exercises — Usual treatment and exercises of cervical mobility before a mirror.
  Arms: Control group
Other: Proprioception exercises — proprioceptive exercises for craniocervical sensorimotor control.
  Arms: Experimental group

SUMMARY:
Introduction: Neck pain is among the most common and costly for industrialized societies. It is difficult to know the exact structure causing the pain so most are considered as non-specific neck pain. There is a correlation between the alteration of craneocervical proprioception and neck pain. The evidence for treatment with proprioceptive exercises is very limited.

Objective: To know the efficacy of a proprioceptive exercise program for neck pain and to compare its effects with a cervical mobility program.

Materials and Methods: Subjects between 18-65 years old with non-traumatic neck pain are included. They will be randomized into two groups of exercises: proprioception or mobility, which will be developed over a period of two weeks, every day, with a total of 10 sessions per patient.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain (NAD I-II) of recent onset (0-3 months)

Exclusion Criteria:

* Cognitive difficulties
* Lack of commitment to attend sessions
* Subjects with pacemakers or defibrillators
* Being receiving another physiotherapeutic treatment
* Other pathologies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Intensity of Pain | four weeks
  Visual Analogue Scale (VAS) was used to register the pain. The VAS is a 10-point rating scale.

SECONDARY OUTCOMES:
Head Repositioning Test | four weeks
  The cervical position is reevaluated with a laser pointer.
Cervical movement range (CROM) | four weeks
  Evaluated with cervical goniometer.
Pain points | four weeks
  Algometer
Neck Disability | four weeks
  Neck Disability Index
Health status | four weeks
  Evaluated with questionnaire of Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Victoria Espí-López, Principal Investigator — fisiotherapy
Locations (1):
- Gemma Victoria Espí-López, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No